CLINICAL TRIAL: NCT03855501
Title: Delayed Apexification Treatment With MTA and Ca(OH)2 of Non-vital Immature Teeth in Adults: A Prospective Comparative Clinical Study
Brief Title: Apexification Treatment With MTA(Mineral Trioxide Aggregate) and Ca(OH)2
Acronym: MTA Ca(OH)2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gözde Kandemir Demirci, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-12/2
Record Dates: First submitted 2019-02-25; First posted 2019-02-26 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Immature Teeth
Keywords: apexification treatment; calcium hydroxide; mineral trioxide aggregate
MeSH Terms: interventions — mineral trioxide aggregate; Calcium Hydroxide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mineral trioxide aggregate (Active Comparator): The root canals were gently instrumented with K-files and copious irrigation was done with 2.5% sodium hypochlorite(NaOCI) by means of a 30 gauge endodontic irrigating needle . After drying with large sterile paper points, calcium hydroxide(CH) paste was mixed with saline and applied to the root canal with a lentulo spiral filler at low speed. A cotton pellet was used to gently compress CH into the root canal and its placement was examined radiographically before placing ZOE as temporary restoration into the access cavity. After one week, CH was removed from the canal by using both the files and the irrigation with 2.5% NaOCI and 17% ethylenediaminetetraacetic acid (EDTA). A final irrigation was made with 2% chlorhexidine (CHX) before obturation. Following drying the root canal with sterile paper points, MTA was placed with a MTA Endo Gun into the apical portion of canals with a minimum 4-mm thickness and adapted to the canal walls with an endodontic hand plugger.
  Interventions: Other: Mineral trioxide aggregate
- Calcium hydroxide (Active Comparator): After using the same biomechanical root canal preparation protocol, the root canal was filled to working length with CH paste. Both clinical and radiographical examinations were performed to evaluate the barrier formation and periapical healing. When a continuous hard tissue barrier was observed apically on radiographs that was verified by clinical probing and complete or significant periapical healing was noticed, the root canal was obturated and coronary restorations were completed as done in MTA group
  Interventions: Other: Calcium hydroxide

INTERVENTIONS:
Other: Mineral trioxide aggregate — Apexification treatment was done with mineral trioxide aggregate
  Arms: Mineral trioxide aggregate
Other: Calcium hydroxide — Apexification treatment was done with calcium hydroxide
  Arms: Calcium hydroxide

SUMMARY:
Ninety immature teeth with necrotic pulps and periapical lesions on patients (aged 16-40y) were treated with AT using MTA (45 teeth) or CH (45 teeth) between 2015 and 2018. The patients were contacted for follow-up examination at 12 to 48 months after treatment. The treatment outcome based on clinical and radiographic criteria was assessed by calibrated examiners and dichotomized as "healed+healing" or "not healed". The age, gender, stage of root development, preoperative signs and symptoms of apical periodontitis and size of periapical lesion were recorded.

DETAILED DESCRIPTION:
The aim of the study was to evaluate and compare the influence of various predictors on outcomes of apexification treatment (AT) using either mineral trioxide aggregate (MTA) or calcium hydroxide (CH) to treat permanent immature anterior teeth with necrotic pulps and periapical lesions in adults. Ninety immature teeth with necrotic pulps and periapical lesions on patients (aged 16-40y) were treated with AT using MTA (45 teeth) or CH (45 teeth) between 2015 and 2018. The patients were contacted for follow-up examination at 12 to 48 months after treatment. The treatment outcome based on clinical and radiographic criteria was assessed by calibrated examiners and dichotomized as "healed+healing" or "not healed". The age, gender, stage of root development, preoperative signs and symptoms of apical periodontitis and size of periapical lesion were recorded. The effect of potential clinical variables on the treatment outcome of AT was evaluated clinically and radiographically during a 12-48-month follow-up. In order to assess the cumulative successes of CH and MTA after AT, Kaplan-Meier survival analysis and log-rank test was used(p>0.05).

ELIGIBILITY:
Inclusion Criteria:

* patients without a systemic disease and compromised immune status
* patients had immature teeth with periapical lesions with or without previous endodontic treatment.

Exclusion Criteria:

* patients with advanced periodontitis (more than 5 mm periodontal attachment and bone loss),
* teeth with contraindications for endodontic treatment (root fracture, unrestorable tooth, replacement resorption or previous surgical endodontic treatment).

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
The rate of the healing of the periapical lesion | 12 to 48 months
  Follow-up visits were performed 12 to 48 months. Changes in apical bone density was evaluated with the modified PAI radiographic healing criteria. The clinical and radiographic healing classification was as follows:
  Healed - the tooth was asymptomatic and the radiograph showed PAI 1 or 2 Healing - the tooth was asymptomatic and the radiograph showed PAI 3 or 4, with score improved at follow up from immediate post-treatment radiograph Not healed - the tooth was either symptomatic or the tooth was asymptomatic but the radiograph presented no decrease or an increase in the size of the pre-existing radiolucency at follow up from immediate post-treatment radiograph (PAI 3-5).
  The treatment outcome was assessed according to the last follow-up data. And all analyses were performed according to the last follow-up data.

CONTACTS AND LOCATIONS:
Overall Officials: Gözde K Demirci, Principal Investigator — Ege University Faculty of Dentistry; Mehmet Emin Kaval, Study Chair — Ege University Faculty of Dentistry; Pelin Güneri, Study Chair — Ege University Faculty of Dentistry; Mehmet Kemal Çalışkan, Study Director — Ege University Faculty of Dentistry

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bonte E, Beslot A, Boukpessi T, Lasfargues JJ. MTA versus Ca(OH)2 in apexification of non-vital immature permanent teeth: a randomized clinical trial comparison. Clin Oral Investig. 2015 Jul;19(6):1381-8. doi: 10.1007/s00784-014-1348-5. Epub 2014 Dec 3. PMID 25467231
- [Result] Damle SG, Bhattal H, Loomba A. Apexification of anterior teeth: a comparative evaluation of mineral trioxide aggregate and calcium hydroxide paste. J Clin Pediatr Dent. 2012 Spring;36(3):263-8. PMID 22838228
- [Result] El-Meligy OA, Avery DR. Comparison of apexification with mineral trioxide aggregate and calcium hydroxide. Pediatr Dent. 2006 May-Jun;28(3):248-53. PMID 16805357